CLINICAL TRIAL: NCT05465343
Title: Efficacy and Safety of Furmonertinib in Patients With EGFR Mutations in Advanced NSCLC With Brain Metastases: A Prospective, Open-label, Phase II Trial（iFORCE）
Brief Title: Furmonertinib in EGFR-Mutant NSCLC With Brain Metastases (iFORCE)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College (Other)
Responsible Party: Principal Investigator, Junling Li, Professor, Peking Union Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC3050
Record Dates: First submitted 2022-07-15; First posted 2022-07-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Furmonertinib; EGFR-mutation; NSCLC; Brain Metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — aflutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- previously treated (Experimental): advanced NSCLC previously treated with systemic therapy, including chemotherapy and targeted therapy
  Interventions: Drug: Furmonertinib 160 mg, Q.D.

INTERVENTIONS:
Drug: Furmonertinib 160 mg, Q.D. — Furmonertinib 160 mg orally once daily in previously treated groups

SUMMARY:
This study is a single-arm, open-label, prospective phase II trial. The aim of this phase II study is to evaluate the efficacy and safety of Furmonertinib in patients with EGFR mutation (including 19del or 21L858R or T790M) in advanced NSCLC with brain metastases.

ELIGIBILITY:
Inclusion Criteria:

1.Male or Female aged ≥18 years old; 2.ECOG PS 0-2; 3.Histologically or cytopathologically confirmed non-small cell lung cancer (NSCLC) ; Tumor tissue samples or blood samples are confirmed to be EGFR mutations (including 19del or 21L858R or T790M); 4.Patients with brain metastases previously treated (chemotherapy, TKI), or intracranial progression after brain radiotherapy； 5.Life expectancy >3 months; 6.Without meningeal metastases; 7.According to mRECIST, the subject has at least 1 intracranial measurable lesion (≥ 5mm); 8.Adequate organ function (28 days before enrollment), including:

1. Blood routine examination HB≥90 g/L（No blood transfusion within 14 days prior to enrollment） ANC≥1.5×109 /L PLT≥100×109 /L
2. Biochemical examination TBIL≤1.5 times ULN AST and ALT≤2.5 times ULN (with liver metastasis, AST and ALT≤5 times ULN) Cr≤1×ULN，CrCL ≥50 mL /min (according to Cockcroft-Gault formula) PT/INR≤1.5 times ULN; aPTT≤1.5 times ULN (If the subject is receiving anticoagulation, PT or aPTT is within the therapeutic range expected for anticoagulant use) 9.No systemic corticosteroid therapy within 4 weeks prior to treatment; 10.Males of reproductive potential or females of potential pregnancy must take effective contraceptive measures (eg, oral contraceptives, intrauterine devices, abstinence or barrier contraception combined with spermicide) during the study and and within 12 months after drug discontinuation; 11.Being able to understand and voluntarily participate in the study, and sign the informed consent form, with good compliance and for follow-up.

Exclusion Criteria:

1.Known or suspected allergy to Furmonertinib or other components; 2.With EGFR Ex20ins mutation; 3.Subjects who have received other anti-tumor therapy within four weeks prior to the first dose of the study or who have failed to recover (≤ grade 1) from an adverse event resulting from prior treatment; 4.Any of the following cardiac criteria:

1. QTc>470 ms on ECG at resting state, when the first abnormality occurs, the test is repeated 2 times within 48h, and the average result of 3 times is calculated.
2. Various clinically significant abnormalities in rhythm, conduction, and resting ECG patterns, such as complete left bundle branch block, third-degree atrioventricular block, second-degree atrioventricular block, PR interval >250msec, etc.
3. Factors that may increase the risk of QTc prolongation or the risk of arrhythmic events.

5.Pregnant or breastfeeding women; 6.Known hepatitis C virus (positive HCV Ab) or human immunodeficiency virus (positive HIV antibody) infection, positive HBsAg or HBCAb with positive HBV DNA copy number (>500 IU/ml); 7.Previous interstitial lung disease (ILD); 8.Having severe or uncontrolled systemic disease, including active opportunistic infection or progressive (severe) infection, uncontrolled diabetes, cardiovascular disease (III or IV heart failure by NYHA Functional Classification, second degree or greater atrioventricular block, myocardial infarction or unstable arrhythmia or unstable angina within the past 6 months, cerebral infarction within 3 months, etc.), pulmonary disease (interstitial pneumonia, obstructive pulmonary disease and history of symptomatic bronchospasm); 9.Meningeal metastases. Intracranial metastases with CNS symptoms may be enrolled if the metastases can be adequately treated and CNS symptoms can be restored to a level less than or equal to CTCAE1 and remain stable prior to enrollment; 10.Received a live vaccination within 4 weeks prior to the start of study treatment; 11.Major surgery (excluding diagnostic surgery) within 4 weeks prior to the start of treatment; 12.Known history of mental disease or drug abuse, and currently having an attack or still taking drugs; 13.Serious gastrointestinal dysfunction, or disease that may affect the intake, transportation or absorption of investigational product; 14.History of other malignant tumors within 3 years, except for cured basal cell carcinoma and cervical carcinoma in situ; 15.According to the investigators, subjects with other serious acute or chronic disease, mental disease , laboratory abnormalities that may increase the risk or interfere with the interpretation of study results are excluded; 16.Subjects who are or have been involved in other clinical studies within 4 weeks; 17.According to the investigator, subjects may not complete this study or may not comply with the requirements of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2025-12-12 (Actual); Study Completion 2025-12-12 (Actual)

PRIMARY OUTCOMES:
Intracranial Progression Free Survival (iPFS) | Approximately 18 months after the first patient begin study treatment
  The time from the first does of the study drugs to the intracranial progression of the disease or death for any reason.

SECONDARY OUTCOMES:
Intracranial Objective Response Rate (iORR) | Approximately 12 weeks after the first patient begin study treatment
  Proportion of subjects whose intracranial tumors were assessed as complete response(CR) or partial response(PR) according to mRECIST.
Intracranial Disease Control Rate (iDCR) | Approximately 18 months from the first patient begin study treatment
  Proportion of subjects whose intracranial tumors were assessed as complete response(CR), partial response(PR), or stable disease(SD) according to mRECIST.
Objective Response Rate (ORR) | Approximately 12 weeks following the first dose of study drug
  Proportion of subjects whose tumors were assessed as complete response(CR) or partial response(PR) according to RECIST 1.1.
Disease Control Rate (DCR) | Approximately 18 months from the first patient begin study treatment
  Proportion of subjects whose tumors were assessed as CR, PR or stable disease (SD) according to RECIST 1.1.
Disease progression free survival (PFS) | Approximately 18 months after the first patient begin study treatment
  The time from the first does of the study drugs to the progression of the disease or death for any reason.
Overall survival (OS) | Approximately 24 months after the first patient begin study treatment
  The time from the first does of the study drugs to the death for any reason.
Adverse Events (AEs) | From the start of study drug to 28 days after the last dose of study drug
  The number of patients with adverse events and the severity according to CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Junling Li, Professor, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Ethics Committee, Beijing, China

IPD SHARING:
Plan to Share IPD: No